CLINICAL TRIAL: NCT00367250
Title: Phase I Study Investigating the Combined Immunotherapy With Trastuzumab and Cetuximab in Patients With Metastatic Breast Cancer With High and Moderate HER2 Expression
Brief Title: Safety Study of Combined Immunotherapy With Trastuzumab and Cetuximab in Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Medical University Vienna, Austria, Dept of Internal Medicine I,
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CETRA 01
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cetuximab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab — weekly i.v.
Drug: Trastuzumab — weekly i.v.

SUMMARY:
One important approach to change the natural history of advanced breast cancer is that of designing new combination chemotherapies in which the best drugs already available are used together with new anticancer agents devoid of clinical cross-resistance. The possibility of exploiting the combined use of cetuximab and trastuzumab represents an option of potential great impact on the probability of response and long-term therapeutic results for patients with advanced breast cancer and HER2 overexpression.Therefore, patients with tumors that demonstrate EGFR expression and clear-cut erbB-2 overexpression (3+) or limited erbB-2 overexpression (+ or 2+) will be included in the study. Patients will be treated with trastuzumab and cetuximab to study the pharmacokinetics and potential drug/drug interaction of both antibodies as well as the safety and tolerability of this novel combination treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of metastatic breast cancer
* presence of at least 1 measurable lesion according to modified RECIST criteria
* Evidence (fluorescence in situ hybridization FISH) of
* Her-2 overexpression in tumor tissue:Group A: Her-2 +++, Group B: Her-2 + or ++
* EGFR-expressing disease as assessed by immunohistochemistry
* Recovered from relevant toxicities from other treatment prior to study entry

Exclusion Criteria:

* Prior treatment with trastuzumab for metastatic breast cancer (adjuvant therapy is allowed)
* Prior treatment with cetuximab
* Concomitant cytotoxic chemotherapy
* Treatment with any investigational agent(s) within 4 weeks prior to study entry
* Known allergic/hypersensitivity reaction to any of the components of study treatments
* severe dyspnea
* Myocardial infarction within 6 months prior to study entry, uncontrolled congestive heart failure; or any current grade 3 or 4 cardio-vascular disorder despite treatment
* History of significant neurologic or psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2006-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics and drug/drug interaction of cetuximab and | repeated PK measurements week 1-13

SECONDARY OUTCOMES:
Safety and tolerability of the combination treatment | week 1 -13
Response | week 9 and 13

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Zielinski, MD, Principal Investigator — Dept of Internal Medicine, Medical University Vienna
Locations (1):
- Dept of Internal Medicine, Vienna, Austria

REFERENCES:
- See also: Dept of Oncology, Medical University Vienna — http://www.meduniwien.ac.at/innere-med-1/onkologie/